CLINICAL TRIAL: NCT03698877
Title: Procalcitonin and Brain Natriuretic Peptides in Patients With Chronic Kidney Disease.
Status: Completed | Type: Observational
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1710018691
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Brain Natriuretic Protein (BNP) and Procalcitonin (PCT) blood tests — For patients with suspected infection, PCT levels will be drawn at the time of suspected infection and again at the start of the next HD treatment.
  For patients with shortness of breath, PCT and BNP levels will be drawn at the time of the complaint and again at the start of the next HD treatment.

SUMMARY:
The study is being conducted to determine if the blood test Brain Natriuretic Protein (BNP) can demonstrate the presence of extra fluid in patients with chronic kidney disease treated by hemodialysis. It will also try to determine the blood test Procalcitonin (PCT) can help identify the cause of the fever, specifically if a fever is caused by a bacterial infection. It will also evaluate whether new blood tests in the future (such as DNA, RNA, metabolite, and protein based tests) can be developed to help predict other complications in patients with chronic kidney disease treated by hemodialysis.

DETAILED DESCRIPTION:
The study has three purposes:

1. To establish a procalcitonin (PCT) algorithm to assist in the identification of bacterial infection in patients with fever and chronic kidney disease (CKD) being treated by hemodialysis;
2. To establish an algorithm to assist clinicians in distinguishing infection from fluid overload in patients with CKD treated by hemodialysis with shortness of breath using PCT and brain natriuretic peptide (BNP);
3. To allow for evaluation of new tests, such as DNA, RNA, metabolite, and protein based tests, which might prove useful in the evaluation of clinical complications encountered by patients with chronic kidney disease treated by hemodialysis including infections and fluid overload.

Baseline Visit:

1. Review of medical and medication history
2. A physical exam and routine clinical laboratory tests (hematology and chemistry) will be performed.
3. PCT and BNP levels will be measured twice prior to hemodialysis (HD) treatment to establish baseline levels.
4. Optional: If the subject consent, samples will be obtained for genetic tests (DNA, RNA, metabolite and proteins) for new tests to be developed in the future.

Follow Up:

1. A physical exam, routine clinical laboratory tests (hematology and chemistry) and medical and medication review will be obtained monthly.

If a subject develops signs of infection or shortness of breath during the course of the study, additional research blood samples for procalcitonin, brain natriuretic peptide, and for genetic testing (Optional) will be obtained as follows:

1. For patients with suspected infection, PCT levels will be drawn at the time of suspected infection and again at the start of the next HD treatment.
2. For patients with shortness of breath, PCT and BNP levels will be drawn at the time of the complaint and again at the start of the next HD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 years and older.
2. Subject is receiving hemodialysis.
3. Able to provide informed consent.

Exclusion Criteria:

1. Subject is unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects are those who are receiving hemodialysis at The Rogosin Institute.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Procalcitonin (ng/mL) | 3 years
  To establish a procalcitonin (PCT) algorithm to assist in the identification of bacterial infection in patients with fever and chronic kidney disease being treated by hemodialysis, PCT levels will be obtained and compared to blood cultures.
Brain Natriuretic Peptide (pg/mL) levels | 3 years
  To distinguish infection from fluid overload, Brain Natriuretic Peptide (BNP) levels will be measured and combined with PCT levels and compared to blood cultures, blood pressure changes and weight (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Silberzweig, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided